CLINICAL TRIAL: NCT03867292
Title: Efficacy of a Physiotherapy Intervention by Electrotherapy Combined With Myofascial Therapy for the Improvement of Lumbar Region Mobility in Federated Padel Players. A Pilot Study
Brief Title: Electrotherapy and Myofascial Therapy in Padel Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MIOTENS
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Low Back Pain, Mechanical
Keywords: Paddle-tennis; Myofascial release; Electrotherapy; Physiotherapy; Low back; Randomized clinical trial
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial (Experimental): The subjects that include the experimental group will receive an intervention through myofascial therapy of crossed hands and electrotherapy
  Interventions: Other: Myofascial
- Electrotherapy (Active Comparator): The subjects that are included in the experimental group will receive an intervention through electrotherapy
  Interventions: Other: Electrotherapy

INTERVENTIONS:
Other: Myofascial — The aim of the application of the crossed hands technique is to produce a deep fascial release, placing the subject in prone position, while the standing physiotherapist will contact with one hand on the spine at the level of the thoracolumbar hinge and with the other hand on the sacrum, so that the hands are crisscrossed. The crossed hands technique will be performed between 90 seconds and 5 minutes.
  The application of the TENS, will be performed for 10 minutes by means of a device, model Compex in the lumbar area, subjects will receive a TENS application of low frequency (less than 40Hz). The electrode - (black) in proximal position or on the most painful zone. The electrode + (red) will be placed distally.
  Arms: Myofascial
Other: Electrotherapy — The application of the TENS, will be performed for 10 minutes by means of a device, model Compex in the lumbar area, subjects will receive a TENS application of low frequency (less than 40Hz). The electrode - (black) in proximal position or on the most painful zone. The electrode + (red) will be placed distally.
  Arms: Electrotherapy

SUMMARY:
Introduction. The lumbar region is one of the locations with the highest incidence of injuries in the paddle players. The crossed hands myofascial technique is used to release the restrictions of the thoracolumbar fascia, improving its mobility. The electrotherapy technique of TENS consists in the application of a low frequency current for the recovery, capitalization and oxygenation of the muscle, thus improving mobility and pain.

Aim. To evaluate the efficacy of an intervention by electrotherapy combined with myofascial therapy, in the lumbar region, for a mobility improvement in older paddle-tennis federated players.

Study design. Randomized, multicenter, simple blind, clinical trial with follow-up period.

Methods. 30 players paddle will be assigned to the two study groups: experimental (intervention through therapy myofascial and electrotherapy) and control (intervention by electrotherapy). The intervention will have a duration of 4 weeks, with 2 sessions per week, lasting 15 minutes. There will be three evaluations: pre-intervention, post-intervention and follow-up. The variable of study is the mobility of the lumbar spine in the movements of flexion and extension (assessed by the employment of tests of Schober and Fingertip-to-floor). The analysis of normality be performed with the Kolmogorov-Smirnof, and in case of homogeneity of the groups is used in parametric tests: test t-student for paired data (difference between the different assessments) and ANOVA of mean repeated (intra-and intersujeto).

Expected results. Improvement of the mobility of the lumbar spine in the movements of flexion and extension.

ELIGIBILITY:
Inclusion Criteria:

* Padel players
* With federal sheet
* Male
* Over 18 years
* Currently participate in regional and / or national competitions

Exclusion Criteria:

* Present a medical diagnosis of musculoskeletal pathology
* Not signed the informed consent document.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline low back flexion after treatment and at a month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Low back flexion will be measured with the Schober test. The subject will remain standing and the evaluator will mark an imaginary line that connects both posterior superior iliac spines (near the Venus pits). A second mark will be placed 10 cm above the first mark and, finally, we will make a third mark 5 cm below the first mark. Next, the subject will be asked to bend to the maximum, keeping the knees extended. When the maximum flexion is reached, the increase in the distance between the skin marks will be measured. The unit of measurement is the centimeter (the greater the distance, the greater the mobility in the flexion of the lumbar spine).

SECONDARY OUTCOMES:
Change from baseline low back extension after treatment and at a month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Low back extension will be measured with the Schober test. The subject will remain standing and the evaluator will mark an imaginary line that connects both posterior superior iliac spines (near the Venus pits). A second mark will be placed 10 cm above the first mark and, finally, we will make a third mark 5 cm below the first mark. Next, the subject will be asked to lean back to the maximum, keeping the knees extended. When the maximum extension is reached, the decrease in the distance between the skin marks will be measured. The unit of measurement is the centimeter (at a lower distance, greater mobility in extension of the lumbar spine).
Change from baseline low back flexion after treatment and at a month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Low back flexion will be measured with the Fingertip-to-floor test. With the subject standing on a platform 20 cm high (without shoes and with their feet together), you will be asked to lean towards flexion, while keeping your knees, arms and fingers fully extended. The vertical distance between the tip of the middle finger and the platform shall be measured with a flexible measuring tape and expressed in centimeters. The vertical distance (measured in centimeters) between the platform and the tip of the middle finger will be positive when the subject does not reach the platform and negative when it can go further.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain